CLINICAL TRIAL: NCT07121712
Title: Efficacy and Neural Mechanisms of Navigated Continuous Theta Burst Stimulation (cTBS) for Generalized Anxiety Disorder (GAD)
Brief Title: Navigated cTBS for the Treatment of Generalized Anxiety Disorder
Acronym: NAVI-GAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WANG KAI (Other)
Responsible Party: Sponsor-Investigator, WANG KAI, Prof., Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AnHuiMU-GAD-cTBS-2025
Record Dates: First submitted 2025-06-29; First posted 2025-08-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Continuous Theta Burst Stimulation; Transcranial Magnetic Stimulation; Neuronavigation; Magnetic Resonance Imaging
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Navigated cTBS (Experimental): Participants will receive active continuous Theta Burst Stimulation (cTBS) guided by a neuronavigation system to the left auditory association cortex. Treatment will be administered three times a day for seven consecutive days.
  Interventions: Device: Mapsd Continuous Theta Burst Stimulation
- Sham Comparator: Sham cTBS (Sham Comparator): Participants will undergo a sham cTBS procedure using a placebo coil that mimics the sound and sensation of the active stimulation but delivers no effective magnetic field. The procedure, including targeting and duration, is identical to the active group to maintain blinding.
  Interventions: Device: Sham Navigated Continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Mapsd Continuous Theta Burst Stimulation — A non-invasive brain stimulation technique using a MagStim Rapid2 stimulator with a 70mm air-cooled figure-of-eight coil. The stimulation target is the left auditory association cortex (MNI: -62, -40, 10), located using a Brainsight neuronavigation system. The cTBS protocol consists of 3-pulse 50 Hz bursts repeated at a 5 Hz frequency for a total of 600 pulses, delivered at 100% of the individual's resting motor threshold (RMT).
  Arms: Experimental: Navigated cTBS
Device: Sham Navigated Continuous Theta Burst Stimulation — A placebo procedure using an inert sham coil that is identical in appearance and sound to the active coil but does not deliver a significant magnetic field to the cortex. All other aspects of the procedure, including neuronavigation, coil placement, duration, and sound, are identical to the active intervention to maintain the blind.
  Arms: Sham Comparator: Sham cTBS

SUMMARY:
The purpose of this study is to investigate the effectiveness of a non-invasive brain stimulation technique called continuous Theta Burst Stimulation (cTBS) for treating Generalized Anxiety Disorder (GAD). The researchers will use a neuronavigation system, which acts like a GPS for the brain based on a participant's own MRI scan, to guide the stimulation to a specific target in the brain's auditory association cortex. This area is involved in processing information and may play a role in anxiety.

Participants who enroll will be randomly assigned to one of two groups. One group will receive active cTBS treatment, while the other will receive a sham (placebo) stimulation that feels similar but has no therapeutic effect. The treatment will be given three times a day for seven consecutive days.

Before and after the treatment period, all participants will complete clinical questionnaires to measure their anxiety and related symptoms. They will also undergo Magnetic Resonance Imaging (MRI) scans to help researchers understand how cTBS affects brain activity. A follow-up assessment will be conducted two weeks after the treatment ends to check on symptoms.

DETAILED DESCRIPTION:
This study is a randomized, triple-blind, sham-controlled trial designed to evaluate the efficacy and neural mechanisms of neuronavigation-guided continuous Theta Burst Stimulation (cTBS) in patients with Generalized Anxiety Disorder (GAD).

A total of 40 patients diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) will be recruited from the First and Second Affiliated Hospitals of Anhui Medical University. After providing informed consent, participants will be randomized in a 1:1 ratio to receive either active cTBS or sham cTBS.

The stimulation target is the left auditory association cortex (posterior superior temporal sulcus), with coordinates derived from previous literature (Neri et al., 2024; MNI coordinates: -62, -40, 10). The TMStarget software will be used to transform these coordinates into each participant's native brain space, and a Brainsight neuronavigation system will guide coil placement for precise targeting.

The active intervention will be delivered using a MagStim Rapid2 stimulator with a 70mm air-cooled figure-of-eight coil. Stimulation intensity will be set at 100% of the individual's resting motor threshold (RMT). The cTBS protocol consists of 3-pulse bursts at 50 Hz, repeated at a 5 Hz frequency, for a total of 600 pulses per session (duration of approximately 41 seconds). The sham intervention will utilize an identical-looking sham coil that produces similar sounds without inducing a significant magnetic field, ensuring the integrity of the blinding.

The treatment schedule consists of three sessions per day, with a 15-minute interval between sessions, for seven consecutive days (from Day 2 to Day 8 of the study protocol).

All participants will undergo comprehensive assessments at baseline (Day 1) and immediately after the final treatment session (Day 9). Assessments include a battery of clinical scales and multimodal magnetic resonance imaging (MRI). The MRI protocol includes high-resolution structural (3D-T1), resting-state functional MRI (rs-fMRI), Diffusion Tensor Imaging (DTI), and specific sequences targeting the Locus Coeruleus. A follow-up assessment of clinical symptoms will be conducted two weeks after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Generalized Anxiety Disorder (GAD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), confirmed by at least two psychiatrists.
2. Hamilton Anxiety Rating Scale (HAMA) score > 14.
3. Age between 18 and 60 years.
4. More than 5 years of education.
5. Right-handed.
6. Normal or corrected-to-normal visual acuity.
7. Able to cooperate with the completion of all experimental procedures.
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Presence of other psychiatric disorders, such as substance abuse, schizophrenia, schizoaffective disorder, hysteria, or autism.
2. Presence of severe neurological diseases (e.g., stroke), or any personal or family history of epilepsy or seizures.
3. Presence of severe somatic diseases, such as severe heart, liver, or renal insufficiency.
4. Pregnant or lactating women.
5. Contraindications to Transcranial Magnetic Stimulation (TMS) or Magnetic Resonance Imaging (MRI), such as the presence of a cardiac pacemaker, cochlear implant, cerebrovascular metal stent, or metal dentures.
6. Inability to cooperate with experimental procedures due to conditions such as depressive stupor or severe claustrophobia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Anxiety Rating Scale (HAMA) Score | Baseline (Day 1), Post-intervention (Day 9), and a 2-week follow-up.
  The HAMA is a 14-item, clinician-administered scale used to assess the severity of anxiety symptoms. Total scores range from 0 to 56, with higher scores indicating more severe anxiety. The change in total score from baseline to post-intervention will be
Change from Baseline in Self-Rating Anxiety Scale (SAS) Score | Baseline (Day 1), Post-intervention (Day 9), and a 2-week follow-up.
  The SAS is a 20-item self-report scale designed to measure the severity of anxiety symptoms. The standard score ranges from 25 to 100, where higher scores indicate more severe levels of anxiety. The change in standard score from baseline will be assessed.
Change from Baseline in Resting-State Neural Activity | Baseline (Day 1) and Post-intervention (Day 9).
  Changes in resting-state brain activity will be measured by functional magnetic resonance imaging (fMRI). Analyses will examine neural activity and network dynamics related to the stimulation target (left auditory cortex) and brain circuits implicated in anxiety.

SECONDARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale (HAMD-17) Score | Baseline (Day 1) and Post-intervention (Day 9).
  The HAMD-17 is a 17-item, clinician-rated scale to assess the severity of depression. Total scores range from 0 to 52, with higher scores indicating more severe depression.
Change from Baseline in Patient Health Questionnaire-15 (PHQ-15) Score | Baseline (Day 1) and Post-intervention (Day 9).
  The PHQ-15 is a 15-item self-report scale to assess the severity of somatic symptoms. Total scores range from 0 to 30, with higher scores indicating more severe somatic symptoms.
Change from Baseline in Four-Dimensional Symptom Questionnaire (4DSQ) Somatization Subscale Score | Baseline (Day 1) and Post-intervention (Day 9).
  The 4DSQ Somatization subscale is a 16-item self-report measure to assess distress from physical symptoms. Scores range from 0 to 32, with higher scores reflecting greater distress from somatization.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Score | Baseline (Day 1) and Post-intervention (Day 9).
  The PSQI is a self-report questionnaire assessing sleep quality. The global score ranges from 0 to 21, with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ji GJ, Ren C, Li Y, Sun J, Liu T, Gao Y, Xue D, Shen L, Cheng W, Zhu C, Tian Y, Hu P, Chen X, Wang K. Regional and network properties of white matter function in Parkinson's disease. Hum Brain Mapp. 2019 Mar;40(4):1253-1263. doi: 10.1002/hbm.24444. Epub 2018 Nov 10. PMID 30414340
- [Background] Neri F, Cappello C, Viberti F, Donniacuo A, Burzi L, Cinti A, Benelli A, Luca Smeralda C, Romanella S, Santarnecchi E, Mandala M, Rossi S. rTMS of the auditory association cortex improves speech intelligibility in patients with sensorineural hearing loss. Clin Neurophysiol. 2024 Apr;160:38-46. doi: 10.1016/j.clinph.2024.02.007. Epub 2024 Feb 9. PMID 38395005